CLINICAL TRIAL: NCT06420297
Title: A Long-term, Open-label Extension Study of Carbetocin Nasal Spray for the Treatment of Hyperphagia in Prader-Willi Syndrome
Brief Title: OLE Study of Carbetocin Nasal Spray for the Treatment of Hyperphagia in Prader-Willi Syndrome
Status: Enrolling by invitation | Phase: Phase 3 | Type: Interventional
Sponsor: ACADIA Pharmaceuticals Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ACP-101-303; 2023-506201-19-00 (EU CTIS Number)
Record Dates: First submitted 2024-05-07; First posted 2024-05-20 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-12

CONDITIONS: Hyperphagia in Prader-Willi Syndrome
Keywords: Opel-label extension; safety; tolerability
MeSH Terms: interventions — carbetocin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Drug: Carbetocin (Experimental): Carbetocin nasal spray 3.2 mg three times daily (TID)
  Interventions: Drug: Carbetocin

INTERVENTIONS:
Drug: Carbetocin — Carbetocin nasal spray 3.2 mg three times daily (TID)
  Other Names: ACP-101

SUMMARY:
To evaluate long-term safety and tolerability of carbetocin nasal spray (3.2 mg TID) in subjects with PWS

DETAILED DESCRIPTION:
This is a long-term, OLE study to evaluate long-term safety and tolerability of carbetocin nasal spray (3.2 mg TID) in subjects with PWS. Subjects who complete the antecedent double-blind study (ACP-101-302) will be invited to participate in the present study.

ELIGIBILITY:
Inclusion Criteria:

* Has completed the Week12/EOT visit of the antecedent, Study ACP-101-302
* Met all entry criteria for the antecedent study
* May benefit from long-term treatment with open-label carbetocin in the judgment of the Investigator.
* Lives with a caregiver who understands and is willing and able to adhere to study-related procedures and is willing to participate in all study visits.

Exclusion Criteria:

* History of, or current, cerebrovascular disease, brain trauma, epilepsy, or frequent migraines. A history of febrile seizures is not exclusionary.
* Active psychotic symptoms, a history of psychotic symptoms, or a psychotic disorder
* History of suicide attempt or inpatient psychiatric hospitalization
* Has a clinically significant abnormality in vital signs at Baseline
* Has an average QTcF interval of >450 ms on the Baseline ECG performed before the first dose of carbetocin is given in the present study (i.e., the ECG performed at the EOT visit of the antecedent study)
* Has developed a clinically significant ECG finding during the antecedent study
* Subject is judged by the Investigator or the Medical Monitor to be inappropriate for the study due to AEs, medical condition, or noncompliance with investigational product or study procedures in the antecedent study

Additional inclusion/exclusion criteria apply. Subjects will be evaluated at screening to ensure that all criteria for study participation are met.

Ages: 5 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 160 (Estimated)
Dates: Start 2024-03-11 (Actual); Primary Completion 2029-05 (Estimated); Study Completion 2029-06 (Estimated)

PRIMARY OUTCOMES:
Treatment-emergent adverse events (TEAEs), serious adverse events (SAEs), withdrawals due to adverse events (AEs), potentially clinically important changes in other safety assessments, device incidents or device malfunctions | Baseline to 36 months
  Treatment-emergent adverse events (TEAEs) and device incidents or device malfunctions, TEAEs leading to discontinuation, TEAEs related to study drug, TEAEs by maximum severity, fatal TEAEs, treatment-emergent SAEs, and treatment-emergent SAEs related to study drug will all be summarized for all subjects as well as by previous treatment group.

CONTACTS AND LOCATIONS:
Locations (30):
- United States (19):
  - Children's of Alabama, Birmingham, Alabama
  - Phoenix Children's Hospital, Phoenix, Arizona
  - University of California Irvine, Orange, California
  - Stanford University School of Medicine, Palo Alto, California
  - Rady Children's Hospital San Diego, San Diego, California
  - Children's Hospital Colorado, Aurora, Colorado
  - Ann & Robert H. Lurie Children's Hospital of Chicago, Chicago, Illinois
  - University of Iowa, Iowa City, Iowa
  - Boston Children's Hospital, Boston, Massachusetts
  - Children's Mercy Kansas City, Kansas City, Missouri
  - SSM Health/Saint Louis University, St Louis, Missouri
  - Maimonides Medical Center, Brooklyn, New York
  - Nationwide Children's Hospital, Columbus, Ohio
  - UPMC-Children's Hospital Pittsburgh, Pittsburgh, Pennsylvania
  - Vanderbilt Clinical Research Center, Nashville, Tennessee
  - Cook Children's Health Care System, Fort Worth, Texas
  - Christus Children's, San Antonio, Texas
  - University of Utah, Salt Lake City, Utah
  - Seattle Children's Hospital, Seattle, Washington
- Canada (2):
  - Alberta Diabetes Institute, Edmonton, Alberta
  - CHU Sainte-Justine, Montreal, Quebec
- Centre Hospitalier Universitaire (CHU) de Toulouse - Hopital des Enfants, Toulouse, Cedex 9 Occitanie, France
- Germany (2):
  - KJF Klinik Josefinum gGmbH, Augsburg
  - Universitätsklinikum Essen, Essen
- Spain (3):
  - Parc Taulí Hospital Universitari, Barcelona
  - Hospital General Universitario Gregorio Marañón, Madrid
  - Hospital Regional Universitario de Málaga, Málaga
- United Kingdom (3):
  - University Hospitals Birmingham NHS Foundation Trust - Heartlands Hospital, Birmingham
  - Royal Hospital for Children Glasgow Clinical, Glasgow
  - Barts Health NHS Trust - The Royal London Hospital, London

IPD SHARING:
Plan to Share IPD: No